CLINICAL TRIAL: NCT03276871
Title: Randomized Controlled Trial Comparing Telescopic Dissection vs. Balloon Dissection During Laparoscopic TEP Inguinal Hernia Repair
Brief Title: Telescopic Dissection vs. Balloon Dissection During Laparoscopic TEP Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Rosen, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-1045
Record Dates: First submitted 2017-09-04; First posted 2017-09-08 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Inguinal Hernia
Keywords: Balloon dissection; Telescopic dissection; Inguinal hernia; TEP
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Balloon Dissection (Active Comparator): Patients will undergo laparoscopic TEP inguinal hernia repair and creation of the extraperitoneal space will be performed with a balloon dissection technique using the Spacemaker Balloon Dissector.
  Interventions: Device: Balloon Dissection
- Telescopic Dissection (Experimental): Patients will undergo laparoscopic TEP inguinal hernia repair and creation of the extraperitoneal space will be performed with a telescopic dissection technique.
  Interventions: Procedure: Telescopic Dissection

INTERVENTIONS:
Procedure: Telescopic Dissection — Creation of extraperitoneal space with blunt dissection using the laparoscopic probe
  Arms: Telescopic Dissection
Device: Balloon Dissection — Creation of extraperitoneal space with aid of the disposable Spacemaker balloon dissector
  Other Names: SpaceMaker Balloon Dissector
  Arms: Balloon Dissection

SUMMARY:
The purpose of this study is to determine if the surgical technique for creation of extraperitoneal space during laparoscopic TEP inguinal hernia repair (telescopic dissection or balloon dissection) has an impact on operative times, early postoperative pain scores, surgical complications and rate of hernia recurrence following laparoscopic TEP inguinal hernia repair.

DETAILED DESCRIPTION:
Minimally invasive approaches have been successfully incorporated into the surgical armamentarium of inguinal hernia repair, with proven benefits for decreased postoperative pain and earlier return to work. Laparoscopic inguinal hernia repair is more commonly performed through the transabdominal preperitoneal (TAPP) approach or the totally extraperitoneal (TEP) approach. The TEP approach has been proven to have equivalent recurrence rates, decreased postoperative pain, earlier ambulation and return to work when compared to the open, tension-free repairs. Additionally, when compared to TAPP, the TEP approach has also been associated with decreased postoperative pain, shorter operative times and equivalent rates of postoperative complications and hernia recurrence.

A key step in the TEP procedure is the creation of the extraperitoneal space, which can be performed by two different techniques: telescopic dissection or balloon dissection.Telescopic dissection is the creation of the extraperitoneal space with blunt dissection performed with the laparoscopic probe. Telescopic dissection was initially described in the original paper describing the TEP procedure, in 1992 by Ferzli et al. To date, telescopic dissection is still used in many centers around the globe. In order to facilitate the creation of the initial working space, disposable dissection balloons have been developed and are commercially available. Balloon dissection is now the most commonly used method for creation of the extraperitoneal space for TEP procedure in the United States. A randomized, prospective multicenter study conducted between 1994 and 1997 and published in 2001 by Bringmam and colleagues has compared operative times, conversion rates, postoperative morbidity and time to return to work between patients in which the TEP procedure was performed with or without the balloon dissector. In this study, the use of the balloon was associated with lower conversion rates and statistically, but perhaps not clinically, significantly shorter operative times (9 minutes difference). No difference was seen in postoperative morbidity, recurrence rates or time to return to work between the groups. Of note, the surgeons performing these procedures were still at an early point of their learning curve for the TEP procedure, which might have influenced the results, especially for the group without the balloon.

Low-cost alternatives have been proposed to substitute the commercially available balloon dissector, especially in developing countries where the access to the balloon dissector is restricted. Despite the fact that the TEP procedure has become more popular in the last 15 years, with surgeons being each time more proficient in this operation, there is a paucity of data comparing cost and surgical outcomes among telescopic and balloon dissection.

Furthermore, according to current consensus, the use of a balloon dissector is especially recommended during the learning period when surgeons are still unfamiliar with the preperitoneal anatomy. Especially for expert surgeons, delineation of the inguinal area and dissection in the creation of extraperitoneal space can be performed as safe and efficient with telescopic dissection.

The investigator's institution has in its staff, three expert surgeons, with a robust experience in the TEP procedure, performed either telescopic or balloon dissection. To help determine if the use of the balloon dissector is associated with a significant decrease in operative times when compared to telescopic dissection, the investigators aim to conduct a randomized controlled trial using the Americas Hernia Society Quality Collaborative (AHSQC) registry. The AHSQC is a nationwide registry designed to improve the value of hernia care using real-time continuous quality improvement principles. Data pertaining to baseline and intraoperative variables, short and long term outcomes are collected prospectively for quality improvement purposes. The information collected in the AHSQC offers a natural repository of information that can be used for research, in addition to its quality improvement purpose.

The investigators hypothesize that at their institution, during TEP repairs, telescopic dissection will be associated with a 15-minute increase in total operative times for a unilateral inguinal hernia, when compared to the balloon dissection.

Specific Aim #1: To determine if the use of a balloon dissector by an experienced surgeon is associated with a significant decrease in total operative time compared to telescopic dissection for the creation of the extraperitoneal space during laparoscopic TEP inguinal hernia repair Specific Aim #2: To determine if there is a difference in postoperative pain scores at 1 day, 7 days and 30 days postoperatively between patients who have undergone laparoscopic TEP inguinal hernia repair performed either with telescopic dissection or balloon dissection.

Specific Aim #3: To determine if there is a difference in the rate of intraoperative complications and 30-day wound events between patients who have undergone laparoscopic TEP inguinal hernia repair performed either with telescopic dissection or balloon dissection.

Specific Aim #4: To determine if 1-year hernia recurrence rates differ between patients who have undergone laparoscopic TEP inguinal hernia repair performed either with telescopic dissection or balloon dissection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent
* Unilateral inguinal hernia
* Scheduled for elective inguinal hernia repair
* Eligible to tolerate general anesthesia
* Eligible to undergo minimally invasive inguinal hernia repair
* Willing to undergo mesh-based repair

Exclusion Criteria:

* Younger than 18 years old
* Unable to give informed consent
* Bilateral Inguinal hernias
* Emergent inguinal hernia repairs ( acute incarceration or strangulation)
* Recurrent inguinal hernia with prior preperitoneal mesh
* Unable to tolerate general anesthesia
* Not eligible for minimally invasive inguinal hernia repair
* Not willing to undergo mesh-based repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rosen, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Comprehensive Hernia Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, rather the results of the aggregate groups of patients will be shared

REFERENCES:
- [Background] Berney CR. Guidelines for laparoscopic (TAPP) and endoscopic (TEP) treatment of inguinal hernia. Surg Endosc. 2012 Nov;26(11):3350-1. doi: 10.1007/s00464-012-2293-5. Epub 2012 Apr 27. No abstract available. PMID 22538696
- [Background] Ferzli GS, Massad A, Albert P. Extraperitoneal endoscopic inguinal hernia repair. J Laparoendosc Surg. 1992 Dec;2(6):281-6. doi: 10.1089/lps.1992.2.281. PMID 1489992
- [Background] Bringman S, Ek A, Haglind E, Heikkinen T, Kald A, Kylberg F, Ramel S, Wallon C, Anderberg B. Is a dissection balloon beneficial in totally extraperitoneal endoscopic hernioplasty (TEP)? A randomized prospective multicenter study. Surg Endosc. 2001 Mar;15(3):266-70. doi: 10.1007/s004640000367. Epub 2001 Feb 27. PMID 11344426
- [Background] Poulose BK, Roll S, Murphy JW, Matthews BD, Todd Heniford B, Voeller G, Hope WW, Goldblatt MI, Adrales GL, Rosen MJ. Design and implementation of the Americas Hernia Society Quality Collaborative (AHSQC): improving value in hernia care. Hernia. 2016 Apr;20(2):177-89. doi: 10.1007/s10029-016-1477-7. Epub 2016 Mar 2. PMID 26936373
- [Derived] Tastaldi L, Bencsath K, Alaedeen D, Rosenblatt S, Alkhatib H, Tu C, Fafaj A, Krpata DM, Prabhu AS, Petro CC, Rosen MJ. Telescopic dissection versus balloon dissection for laparoscopic totally extraperitoneal inguinal hernia repair (TEP): a registry-based randomized controlled trial. Hernia. 2019 Dec;23(6):1105-1113. doi: 10.1007/s10029-019-02001-y. Epub 2019 Aug 6. PMID 31388790

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Balloon Dissection | Telescopic Dissection
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balloon Dissection | Telescopic Dissection | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 10 | 26
  >=65 years | 5 | 9 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 20 | 16 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 26 [24.3 to 27.5] | 25.7 [24.4 to 28.9] | 25.9 [24.2 to 27.8]
Diabetes [Count of Participants; unit: Participants] | 0 | 2 | 2
Smoking [Count of Participants; unit: Participants] | 5 | 2 | 7
COPD [Count of Participants; unit: Participants] | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: Total Operative time measured in minutes, from incision to end of procedure; operative times will be reported as median and interquartile range.
Time Frame: Measured from start to end of procedure
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Balloon Dissection | Telescopic Dissection
Number analyzed (Participants) | 21 | 19
minutes | 46 [33 to 63] | 43 [35 to 90]

2. Secondary Outcome: NRS-11 Pain Scores
Description: Early postoperative pain scores; Pain scores measured with the Numeric Pain Rating Scale (NRS-11) pain score at postoperative days 1, 7 and 30. Pain ratings will be reported as median and inter-quartile range. Scores can range from 0 to 10, higher numbers represent more pain.
Time Frame: Postoperative day 1, Postoperative day 7 and Postoperative day 30
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Balloon Dissection | Telescopic Dissection
Number analyzed (Participants) | 21 | 19
units on a scale
  NRS-11, Postop day 1 | 3 [2 to 4] | 4 [3 to 5]
  NRS-11, Postop day 7 | 2 [0.75 to 3.25] | 1.5 [0.25 to 3.0]
  NRS-11, 30-day | 0.5 [0 to 2] | 0 [0 to 2.75]

3. Secondary Outcome: Number of Participants With Intra-operative Complications
Description: Rate of any Intra-operative complications; rate will be reported in number and percent as appropriate
Time Frame: Intraoperative complications recorded during the procedure, up to closure of the incisions
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Dissection | Telescopic Dissection
Number analyzed (Participants) | 21 | 19
Participants | 1 | 0

4. Secondary Outcome: 30-day SSO (Surgical Site Occurrences) Rate
Description: 30-day rate of Surgical Site Occurrences which includes any surgical site infection as well as wound cellulitis, non-healing incisional wound, fascial disruption, skin or soft tissue ischemia, skin or soft tissue necrosis, wound serous drainage, seroma, hematoma, or development of an enterocutaneous fistula. The rate will be reported in number and percent as appropriate
Time Frame: 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Dissection | Telescopic Dissection
Number analyzed (Participants) | 21 | 19
Participants | 4 | 0

ADVERSE EVENTS:
Time Frame: The adverse event data were collected up to 30 days following surgery
Arm/Group | Balloon Dissection | Telescopic Dissection
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/19
Other Adverse Events (participants affected / at risk) | 0/21 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Dissection (N=21) | Telescopic Dissection (N=19)
Port site hernia requiring reoperation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Dissection (N=21) | Telescopic Dissection (N=19)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03276871/Prot_SAP_000.pdf